CLINICAL TRIAL: NCT06213727
Title: To Evaluate the Efficacy and Safety of ZKY001 Eye Drops in the Treatment of Corneal Epithelial Defects in a Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ⅱ Clinical Trial
Brief Title: ZKY001 Eye Drops in the Treatment of Corneal Epithelial Defects in a Phase Ⅱ Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKO-SFT-202106-PTY
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Corneal Epithelial Defect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial drug group 1 (Experimental): lowe-dose ZKY001 eye drops
  Interventions: Drug: lowe-dose ZKY001 eye drops
- Trial drug group 2 (Experimental): Medium-dose ZKY001 eye drops
  Interventions: Drug: Medium-dose ZKY001 eye drops
- control group (Placebo Comparator): ZKY001 simulated eye drops
  Interventions: Drug: ZKY001 simulated eye drops

INTERVENTIONS:
Drug: lowe-dose ZKY001 eye drops — eye drops
  Arms: Trial drug group 1
Drug: Medium-dose ZKY001 eye drops — eye drops
  Arms: Trial drug group 2
Drug: ZKY001 simulated eye drops — eye drops
  Arms: control group

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled clinical trial was designed. The study included two experimental groups (low-dose ZKY001 eye drops group and medium-dose ZKY001 eye drops group) and a placebo control group, with 60 subjects in each group.

DETAILED DESCRIPTION:
Each subject had the study drug instilled into the study eye according to the randomly obtained drug number.

Duration OF THE STUDY：The screening period was D-5 to D-1, the experimental period was D0 (the day of operation) to D5, and the observation period was D10±2.

Statistical analyses were performed with the use of SAS software (version 9.4 or higher) without special instructions. All statistical tests were two-sided, with a significance level of 0.05. Enrollment analysis: the number of enrolled and completed cases in each center was summarized, and the list of dropped cases was made. Overall dropout rates in each group and dropout rates related to adverse events were compared between groups with the use of the chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-70 years old, both sexes;
2. patients were diagnosed as primary pterygium with nasal onset, and the head tip of pterygium invaded the cornea ≥3mm and ≤5mm, and underwent pterygium excision combined with conjunctival autotransplantation with autologous limbal stem cells;
3. Except for the pterygium neck under the slit lamp during the screening period, the limbal anatomy was normal without obvious abnormalities (e.g., scar, neovascularization that had invaded the cornea, or pseudopterygium);

Exclusion Criteria:

1. secondary pterygium, recurrent pterygium, pseudopterygium, bilateral pterygium or conjunctival tumor;
2. Schirmer test I (topical anesthesia) ≤3mm/5min;
3. severe blepharitis and/or severe meibomian gland disease, recurrent corneal erosion, chronic corneal disease, chemical burn and other ocular diseases that seriously affect ocular surface structure or function;
4. patients with syphilis, Sjogren's syndrome, cicatricial pemphigoid and other systemic diseases that seriously affect ocular surface structure or function;
5. rheumatoid arthritis, Sjogren syndrome, systemic lupus erythematosus, AIDS and other autoimmune diseases;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Corneal epithelial defect repair area | 3 days
  Percentage improvement of corneal epithelial defect area from baseline in the afternoon of D3

SECONDARY OUTCOMES:
VAS score | 5 days
  the mean change of VAS scores from baseline in D3 and D5
Best Corrected Visual acuity (BCVA) | 5 days
  The mean change of best corrected visual acuity at D1, D3, and D5 from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Shandong First Medical University (Shandong Eye Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No